CLINICAL TRIAL: NCT07236528
Title: A Prospective, Multicenter, Single Arm, Open Label Clinical Study Evaluating the Efficacy and Safety of the Combination of Carilizumab With Apatinib Mesylate and Radiotherapy in the First-line Treatment of Advanced Mucosal Melanoma
Brief Title: Combination of Carilizumab, Apatinib, and Radiotherapy for Advanced Mucosal Melanoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Zhengyun Zou, professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0433-01
Record Dates: First submitted 2025-09-28; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Mucosal Melanoma
Keywords: radiotherapy; Carilizumab; Apatinib Mesylate; Mucosal melanoma; first-line treatment
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of Carilizumab with Apatinib Mesylate and Radiotherapy (Experimental)
  Interventions: Drug: Carilizumab and Apatinib

INTERVENTIONS:
Drug: Carilizumab and Apatinib — Carilizumab 200mg, intravenous infusion, administered once every 2 weeks, with a 4-week cycle; Apatinib mesylate 500mg, oral, once daily, adjusted according to patient tolerance, with a 4-week cycle; Completed 2 cycles in total. ·Synchronous radiotherapy stage: 200mg of Carilizumab is administered intravenously once every 2 weeks, with a 4-week cycle; Apatinib mesylate 500mg, oral, once daily, adjusted according to patient tolerance, with a 4-week cycle;

SUMMARY:
This study is a prospective, multicenter, single arm, open label study aimed at evaluating the efficacy and safety of the combination of Carilizumab, Apatinib Mesylate, and first-line radiotherapy for advanced mucosal melanoma.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single arm, open label study aimed at evaluating the efficacy and safety of the combination of Carilizumab, Apatinib Mesylate, and first-line radiotherapy for advanced mucosal melanoma. The study will use the 6-month progression free survival rate (PFS6) as the primary efficacy indicator and plan to enroll approximately 30 non-surgical first-line treatment subjects with mucosal melanoma. After being fully informed and signing informed consent forms, the subjects will be screened and qualified to receive the following treatments: Induction phase (2 cycles): 200mg of Carilizumab, intravenous infusion, administered once every 2 weeks, with a 4-week cycle; Apatinib mesylate 500mg, oral, once daily, adjusted according to patient tolerance, with a 4-week cycle; Completed 2 cycles in total. ·Synchronous radiotherapy stage: 200mg of Carilizumab is administered intravenously once every 2 weeks, with a 4-week cycle; Apatinib mesylate 500mg, oral, once daily, adjusted according to patient tolerance, with a 4-week cycle; The radiation therapy plan evaluated by the researchers: the radiation dose and radiation field are determined by the researchers, with an overall principle of 18-25Gy/3-6f, or equivalent BED. Three dimensional conformal radiotherapy (3D-CRT) or intensity-modulated conformal radiotherapy (IMRT) techniques are used for radiotherapy. Radiotherapy should be scheduled before the use of PD-1 antibody Carilizumab, and intravenous infusion of Carilizumab should be administered within 48 hours after the end of radiotherapy. If there are multiple lesions that can be treated with radiotherapy, after evaluation by the research team, sequential radiotherapy for multiple lesions is allowed based on the lesion location and the tolerance of surrounding normal organs. ·Maintenance phase: Carilizumab 200mg, intravenous infusion, administered once every 2 weeks, with a 4-week cycle; Apatinib mesylate 500mg, oral, once daily, adjusted according to patient tolerance, with a 4-week cycle; Until tumor progression, intolerance, initiation of other anti-tumor treatments, loss to follow-up, or death. The cumulative maximum shall not exceed 2 years. After the completion of treatment, subjects will continue to undergo post-treatment safety and survival follow-up. For subjects who have completed treatment due to non disease progression/death reasons, tumor progression follow-up will also be conducted after the completion of treatment. Safety visit: After the subjects are enrolled in the study, safety visits will be conducted at each treatment cycle D1 and at the end of treatment visit. Imaging assessment: All lesions were recorded and evaluated according to RECIST 1.1. The window period allowed for imaging examinations is ± 7 days unless otherwise specified. During the research period, unplanned imaging examinations may be performed when tumor progression is suspected. The assessment of tumor baseline within 4 weeks before enrollment, CT/MRI scan results obtained before signing informed consent can be used for screening tumor assessment as long as they meet the requirements; Suspected brain metastases require enhanced MRI/CT of the brain to rule out brain metastases. When there is a clear or clinical suspicion of bone metastasis, bone scan examination should be performed to exclude bone metastasis. Within 12 months after the first administration, imaging examinations should be conducted every 2 cycles (± 7 days). After 12 months, imaging examinations should be conducted every 3 cycles (± 7 days). If there is suspicion of metastasis to other areas, additional imaging examinations for that area should be performed. After terminating the study treatment, subjects who did not show imaging progression continued to undergo imaging evaluation at the frequency of the treatment period until imaging progression, acceptance of other anti-tumor treatments, withdrawal of informed consent, loss to follow-up, or death occurred. Survival follow-up: After the completion or withdrawal of the study, survival and post study information will be collected through telephone follow-up every 3 months until death, loss to follow-up, withdrawal of informed consent, observation for 1 year, or termination of the study by the researcher.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 80 years old, gender not limited
2. Confirmed by pathological histology, patients with recurrent, unresectable, or metastatic mucosal melanoma after surgery
3. In the late stage, no systemic anti-tumor drug treatment has been received, and previous radical surgical resection, adjuvant or neoadjuvant therapy is allowed. However, it is required to be completed at least 4 weeks before randomization, and all treatment-related toxicity events have returned to normal or CTCAE 5.0 grade I or below (except for hair loss, skin hypopigmentation, well controlled hypothyroidism, and adrenal insufficiency)
4. There must be at least one measurable lesion that has not undergone local treatment (according to RECIST v1.1 requirements, the length of the measurable lesion on spiral CT or MRI scan must be ≥ 10 mm or the length of enlarged lymph nodes must be ≥ 15 mm)
5. At least one lesion that can receive radiotherapy
6. ECOG PS 0 or 1 point
7. Expected survival period ≥ 12 weeks
8. No contraindications for treatment, with sufficient organ and bone marrow function: ① Absolute neutrophil count ≥ 1.5 × 109/L ② Platelets ≥ 80 × 109/L③ Hemoglobin ≥ 90 g/L④ ALT and AST ≤ 1.5 × ULN⑤ Bilirubin ≤ 1.5 × ULN⑥ Blood creatinine ≤ 1.5 × ULN
9. Patients may have a history of brain/meningeal metastases, but they must have undergone local treatment (surgery/radiation therapy) before the start of the study and have been clinically stable for at least 3 months (corticosteroids are allowed to be used before randomization, but must be discontinued 2 weeks before starting the study drug)
10. Non surgical sterilization or female patients of childbearing age are required to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill, or condom) during the study treatment period and within 12 months after the end of the study treatment period
11. For male patients whose partners are women of childbearing age, effective contraception methods should be used during the trial period and within 12 months after the last dose. 11. Participants voluntarily join the study, sign informed consent forms, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Patients who have received VEGFR TKI treatment within the past 6 months (including neoadjuvant and adjuvant treatment periods)
2. Individuals known to be allergic to recombinant humanized anti-PD-1 monoclonal antibody drugs and their components
3. History of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation
4. Previous thyroid dysfunction and inability to maintain normal thyroid function even with medication treatment
5. Pregnant or lactating women
6. Evidence of bleeding quality or significant coagulation dysfunction (not receiving anticoagulant therapy)
7. Bleeding events occurring within 6 months prior to the first medication due to untreated or incompletely treated esophageal and/or gastric varices
8. Major vascular disease (such as aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) occurred within 6 months before the first use of medication
9. Insufficient control of hypertension (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90mmHg) (based on the average of BP readings obtained from ≥ 2 measurements), allowing for the use of antihypertensive therapy to achieve the above parameters
10. Previously experienced hypertensive crisis or hypertensive encephalopathy
11. Within the past 3 months, there has been severe cardiovascular disease (such as New York Heart Association Grade II or above heart disease, myocardial infarction, or cerebrovascular accident), unstable arrhythmia, or unstable angina pectoris
12. Severe, unhealed, or cracked wounds, active ulcers, or untreated fractures
13. Perform hollow needle biopsy or other minor surgery within 3 days before the first medication, excluding the placement of vascular access devices
14. Major surgery should be performed within 4 weeks before the first medication, or expected to be required during the study period
15. Those who have been treated with systemic immunosuppressive drugs (including but not limited to glucocorticoids [>10 mg/d prednisone or other corticosteroids with equivalent physiological doses], cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor alpha [TNF - α] preparations) within 2 weeks prior to their first medication, or who are expected to require systemic immunosuppressive drugs during the study treatment period
16. Subjects who have received or will receive a live vaccine within 30 days prior to the first dose, or who are expected to use the vaccine during the expected treatment period or within 5 months after the last dose

176. Individuals known to be allergic to any investigational drug or excipient

18. Individuals with a history of abuse of psychotropic drugs who are unable to quit or have mental disorders

19. Researchers determine other situations that are not suitable for inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
6-month progression free survival rate | From the day each patient starts treatment until the 6th month (180 days).

SECONDARY OUTCOMES:
Overall survival, OS | every 3 months after the patient completed the trial treatment
Disease control rate,DCR | The subjects must be confirmed at least 4 weeks ± 7 days after the initial evaluation.
objective response rate | The subjects must be confirmed at least 4 weeks ± 7 days after the initial evaluation.

IPD SHARING:
Plan to Share IPD: No